CLINICAL TRIAL: NCT01823991
Title: Pilot Clinical Trial of COGNUTRIN in Breast Cancer Survivors
Brief Title: COGNUTRIN in Breast Cancer Survivors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Gateway for Cancer Research (Other); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MCC-17089
Record Dates: First submitted 2013-04-01; First posted 2013-04-04 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: polyphenolics; anthocyanins; n-3 fatty acids
MeSH Terms: conditions — Breast Neoplasms | interventions — blueberry extract; Anthocyanins; Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COGNUTRIN (VITABLUE and n-3 fatty acids) (Experimental): Participants will be provided with two bottles containing Lovaza and VitaBlue. Participants will be asked to take 1 tablet of Lovaza two times a day and 1 tablet of VitaBlue three times a day.
  Interventions: Drug: VitaBlue™; Drug: Lovaza®
- Placebo Administration (Placebo Comparator): Participants will be provided with two bottles containing placebo. Participants will be asked to take 1 tablet of one placebo two times a day and 1 tablet of other placebo three times a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VitaBlue™ — Self administration of nutritional supplement COGNUTRIN for 3 months.
  The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.
  Other Names: blueberry (BB) Anthocyanins
  Arms: COGNUTRIN (VITABLUE and n-3 fatty acids)
Other: Placebo — Self administration of placebo for 3 months.
  Investigators use a placebo to make sure that it really is the study medicine that is making a difference in the participant's condition. It does not have anything in it that would normally help or harm most people.
  Arms: Placebo Administration
Drug: Lovaza® — Self administration of nutritional supplement COGNUTRIN for 3 months.
  The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.
  Other Names: omega-3-acid ethyl esters
  Arms: COGNUTRIN (VITABLUE and n-3 fatty acids)

SUMMARY:
The purpose of this study is to examine the safety and influence of an intervention (COGNUTRIN) using nutritional supplements (n-3 fatty acids and blueberry anthocyanins) on cognitive performance in breast cancer survivors following chemotherapy. The investigators' goal is to treat or lessen the late effects of cancer treatment. The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.

DETAILED DESCRIPTION:
This pilot study will evaluate the feasibility of administration of the nutritional supplement and placebo in this patient population and performing cognitive function testing at baseline and post supplementation.

This is a randomized, double-blind pilot study of COGNUTRIN vs. Placebo.

Participants have an equal chance (like flipping a coin) of being in either of the study groups. Neither the participant nor the study doctor will be able to choose which study group the participant is in. Participants will not know and the study doctor will not know which study group the participants are in.

ELIGIBILITY:
Inclusion Criteria:

* Cases with Stage II-IIIA Breast Cancer that have completed adjuvant treatment with anthracyclines and/or taxanes + or -Radiation therapy within past 6 months(+/- 7 days) (subjects on concurrent endocrine therapy (TAM, Aromatase inhibitors are also eligible to participate as this is standard of care for this patient population)
* Able to understand and sign the informed consent
* Fluent in reading, comprehension and communication in the English language
* No evidence of dementia - Mini Mental State Examination (MMSE) >=23 but some evidence of cognitive impairment
* Must be aware of the nature of his current medical condition and must be willing to give consent after being informed of the experimental nature of therapy, alternatives, potential benefits, side-effects, risks and discomforts
* Eastern Cooperative Oncology Group (ECOG) performance status of 0- 2 (Karnofsky score >60%)
* Acceptable hemoglobin and hematocrit level based on complete blood count (CBC)
* Must be willing to be monitored for adequacy of nutritional intake during the intervention, as is the current standard of clinical practice

Exclusion Criteria:

* Use of estrogens (oral, dermal or vaginal), progesterone (oral or topical), androgens, Raloxifene or Tamoxifen during the previous 3 months
* Use of over the counter steroid hormonal supplements including dehydroepiandrosterone (DHEA)
* Patients with advanced or Stage IIIIB or IV breast cancer or other cancers
* Use of n-3 fatty acids or high dose antioxidant supplements other than what is provided in the trial
* History of known allergy to components of the study supplements
* Renal or liver disease
* Concurrent participation in another chemoprevention trial
* Evidence of bleeding diathesis or coagulopathy
* Metabolic abnormalities (e.g. thyroid disorders, insulin dependent diabetes, rheumatologic disease etc.)
* Known claustrophobia, presence of pacemaker and/or ferromagnetic material in their body that would prohibit MRI imaging
* Medical history of concussions
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or study drug administration, or may interfere with interpretation of study results, and in the judgment of the investigator would make the potential participant inappropriate for entry into this study

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2018-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Kumar, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center between July 2014 and February 2017.
Pre-assignment Details: Participants were randomized to receive Cognutrin (n-3 fatty acids + anthocyanins) or placebo for a period of 3 months.
Groups:
- COGNUTRIN (n-3 Fatty Acids + Anthocynins) Twice a Day (BID): Participants will be provided with two bottles containing Lovaza and VitaBlue. Participants will be asked to take 1 tablet of Lovaza two times a day and 1 tablet of VitaBlue three times a day.
  VitaBlue™: Self administration of nutritional supplement COGNUTRIN for 3 months.
  The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.
  Lovaza®: Self administration of nutritional supplement COGNUTRIN for 3 months.
  The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.
- Matching Placebo BID: Participants will be provided with two bottles containing placebos. Participants will be asked to take 1 tablet of placebo two times a day and 1 tablet of or placebo three times a day.
  Placebo: Self administration of placebo for 3 months.
  Investigators use a placebo to make sure that it really is the study medicine that is making a difference in the participant's condition. It does not have anything in it that would normally help or harm most people.
Period: Overall Study
Arm/Group | COGNUTRIN (n-3 Fatty Acids + Anthocynins) Twice a Day (BID) | Matching Placebo BID
Started | 18 | 18
Completed | 10 | 13
Not Completed | 8 | 5
Not completed — Withdrawal by Subject | 8 | 5

BASELINE CHARACTERISTICS:
Population: All Participants.
Groups:
- COGNUTRIN (n-3 Fatty Acids + Anthocynins) Twice a Day (BID): Participants will be provided with two bottles containing Lovaza (or placebo) and VitaBlue (or placebo). Participants will be asked to take 1 tablet of Lovaza (or placebo) two times a day and 1 tablet of VitaBlue (or placebo) three times a day.
  VitaBlue™: Self administration of nutritional supplement COGNUTRIN for 3 months.
  The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.
  Lovaza®: Self administration of nutritional supplement COGNUTRIN for 3 months.
  The supplement to be used will be a combination of the following: (1) VitaBlue (40% polyphenolics, 12.5% anthocyanins from blueberries (BB) and (2) n-3 fatty acids - Lovaza.
- Matching Placebo BID: Participants will be provided with two bottles containing Lovaza (or placebo) and VitaBlue (or placebo). Participants will be asked to take 1 tablet of Lovaza (or placebo) two times a day and 1 tablet of VitaBlue (or placebo) three times a day.
  Placebo: Self administration of placebo for 3 months.
  Investigators use a placebo to make sure that it really is the study medicine that is making a difference in the participant's condition. It does not have anything in it that would normally help or harm most people.
- Total: Total of all reporting groups
Arm/Group | COGNUTRIN (n-3 Fatty Acids + Anthocynins) Twice a Day (BID) | Matching Placebo BID | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (4.85) | 50.92 (6.17) | 46 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function Scores With Intervention - HVLT and COWA
Description: Mean change in cognitive function scores measured from baseline to post intervention with Cognutrin compared to placebo. Mean cognitive function scores by group and compared by time of testing (Time 1, Time 2). The HVLT test assesses verbal learning and memory. Subjects are given a list of words and asked to repeat as many words as they can recall at 3 times. There is no absolute low & high, as scores are age adjusted. Reported scores are T-scores- average score should be 50, with a standard deviation of 10. Any score below 50 indicates performance below population averages and any score above 50 indicates higher than population averages.The COWA test is a verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with a designed letter. The scores are converted to z-scores. A Z score of -1 is 1 standard deviation below mean. The lowest and highest Z scores could be ≤ -3.0 and ≥3.0. A lower Z score is indicative of poor fluency.
Time Frame: Baseline (Time 1) and at 3 months +/- 7 days (Time 2)
Population: All evaluable participants at time of analysis.
Measure: Mean (Standard Error); unit: score
Groups:
- A - Cognutrin #1: Cognutrin Treatment Time 1
- B - Cognutrin #2: Cognutrin Time 2.
- C - Placebo #1: Placebo Time 1.
- D - Placebo #2: Placebo Time 2.
Arm/Group | A - Cognutrin #1 | B - Cognutrin #2 | C - Placebo #1 | D - Placebo #2
Number analyzed (Participants) | 5 | 5 | 10 | 10
score
  HVLT-total recall | 49.04 (6.41) | 44.93 (7.55) | 42.28 (4.21) | 43.33 (4.96)
  HVLT-delayed recall | 44.82 (5.33) | 41.59 (7.02) | 47.49 (3.5) | 44.1 (4.62)
  COWA-z score | -.341 (.686) | -.452 (.577) | -0.001 (0.451) | 0.332 (0.379)

2. Primary Outcome: Change in Cognitive Function Scores With Intervention - Color Trails 1 & 2
Description: Mean change in cognitive function scores measured from baseline to post intervention with Cognutrin compared to placebo arms of the trial. Mean cognitive function scores by group and compared by time of testing (Time 1, Time 2). Tests: Color Trails 1 & Color Trails 2. Color Trails 1 consists of a page with scattered circles numbered from 1-25. Even numbered circles are colored yellow and odd numbered ones are colored pink. Respondents are instructed to connect the circles in consecutive numeric order with a continuous line as quickly as possible. Score is determined by recording the number of seconds required to complete the task. Color Trails 2 consists of a page containing 25 pink circles and 25 yellow circles numbered 1-60. Respondents are instructed to connect circles in consecutive order while alternating colors. A total score is determined by recording the number of seconds required to compete the task.
Time Frame: Baseline (Time 1) and at 3 months +/- 7 days (Time 2)
Population: All evaluable participants at time of analysis.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | A - Cognutrin #1 | B - Cognutrin #2 | C - Placebo #1 | D - Placebo #2
Number analyzed (Participants) | 4 | 4 | 10 | 10
seconds
  Color Trails 1 | 59.82 (11.5) | 61.25 (4.87) | 47.47 (2.89) | 50.80 (2.76)
  Color Trails 2 | 60.35 (4.35) | 60.57 (4.64) | 54.96 (2.47) | 59.97 (2.63)

3. Primary Outcome: Change in Cognitive Function Scores With Intervention - Digit Span
Description: Mean change in cognitive function scores measured from baseline to post intervention with Cognutrin compared to placebo. Mean cognitive function scores by group and compared by time of testing (Time 1, Time 2). The Digit Span assesses immediate verbal memory and auditory attention. The examiner reads increasingly longer series of numbers and the respondent is required to repeat them in the same order. The examiner then reads additional sequences of numbers and the respondent is required to repeat them in reverse order. Digit Span yields one score, number of items completed correctly. Scores are scaled from the Wechsler Adult Intelligence Scale. The values for these scaled scores indicated that values from 1-7 indicate below average performance, corresponding to 1-16 percentile ranks. Scores between 8-12 indicate average performance, corresponding to percentile ranks of 25-75. Scores between 13-19 correspond to areas of strength and 84-99 percentile ranks.
Time Frame: Baseline (Time 1) and at 3 months +/- 7 days (Time 2)
Population: All evaluable participants at time of analysis.
Measure: Mean (Standard Error); unit: score
Arm/Group | A - Cognutrin #1 | B - Cognutrin #2 | C - Placebo #1 | D - Placebo #2
Number analyzed (Participants) | 5 | 5 | 11 | 11
score | 9.58 (1.43) | 12.69 (1.75) | 10.01 (.89) | 10.05 (1.09)

4. Primary Outcome: Change in Cognitive Function Scores With Intervention - Symbol Digit Modalities Test
Description: Mean change in cognitive function scores measured from baseline to post intervention with Cognutrin compared to placebo arms of the trial. Mean cognitive function scores by group and compared by time of testing (Time 1, Time 2). The Symbol Digit Modalities Test requires respondents to write the number that corresponds with each symbol for a series of 110 items in which the symbol but not the number appears. Respondents identify the correct number using a key provided in which symbols are matched with numbers. Total score is determined by calculating the number of items correctly completed in 90 seconds Scale uses z-scores which have a mean of 0 and a standard deviation of 1. Scores cores above 0 indicate better than average performance whereas scores below 0 indicate poorer than average performance.
Time Frame: Baseline (Time 1) and at 3 months +/- 7 days (Time 2)
Population: All evaluable participants at time of analysis.
Measure: Mean (Standard Error); unit: score
Arm/Group | A - Cognutrin #1 | B - Cognutrin #2 | C - Placebo #1 | D - Placebo #2
Number analyzed (Participants) | 4 | 4 | 11 | 11
score | .17 (.72) | .39 (.62) | .53 (.39) | .72 (.33)

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The primary safety endpoint is incidence and severity of AEs occurring during intervention with either COGNUTRIN or placebo. All AEs that are reported by the participant, detected during a visit, physical examination, or laboratory work-up will be recorded in the participant's medical record and recorded on the case report form (CRF). All AEs that occur after the informed consent is signed will be recorded on the AE CRF whether or not related to study agent, using the NCI Common Terminology Criteria for AEs (CTCAE) version 4.0.
Time Frame: 3 months from baseline +/- 7 days
Population: All evaluable participants who received treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID): Self administration of nutritional supplement COGNUTRIN for 3 months.
- Matching Placebo Twice a Day (BID): Self administration of placebo for 3 months.
Arm/Group | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) | Matching Placebo Twice a Day (BID)
Number analyzed (Participants) | 16 | 16
Participants | 10 | 4

6. Secondary Outcome: Occurrence of Adverse Events (AEs) by Causality
Description: Number of Adverse events according to relation to study treatment category: Definitely related, Probably related, Possibly related, Unlikely to be related, Unrelated.
Time Frame: 3 months from baseline +/- 7 days
Population: Participants with Adverse Events.
Measure: Number; unit: Adverse Events
Arm/Group | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) | Matching Placebo Twice a Day (BID)
Number analyzed (Participants) | 10 | 4
Adverse Events
  Definitely related to treatment | 5 | 0
  Probably related to treatment | 1 | 0
  Possibly related to treatment | 0 | 0
  Unlikely to be related to treatment | 0 | 0
  Unrelated to treatment | 11 | 8

7. Secondary Outcome: Number of Participants Experiencing Grade 3 or Higher Adverse Events
Description: The primary safety endpoint is incidence and severity of AEs occurring during intervention with either COGNUTRIN or placebo. All AEs that are reported by the subject, detected during a visit, physical examination, or laboratory work-up will be recorded in the participant's medical record and recorded on the case report form (CRF). All AEs that occur after the informed consent is signed will be recorded on the AE CRF whether or not related to study agent, using the NCI Common Terminology Criteria for AEs (CTCAE) version 4.0.
Time Frame: 3 months from baseline +/- 7 days
Population: Evaluable participants who received treatment.
Measure: Number; unit: participants
Arm/Group | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) | Matching Placebo Twice a Day (BID)
Number analyzed (Participants) | 16 | 16
participants | 0 | 0

8. Secondary Outcome: Number of Participants With Improvement in Function MRI and Structural MRI Post-Intervention
Description: Functional: Improved cortical activation in multiple areas of the brain on examination of functional MRI post study intervention. Imaging including: 1) Extended resting state functional MRI with data post-processed on Philips EWS. Performed with patient's eyes closed and minds wandering. 2) Diffusion tensor imaging (DTI) with effective slice thickness of 2.3mm. Post-processed on Philips EWS with color-coded DTI tractography images obtained, absolute FA calculations performed in 9 anatomic areas in both right and left brain with total of 18 FA values obtained per examination. Structural: Improved white matter signal changes which correlate with ischemic changes or microvascular ischemic changes, cortical atrophy, hippocampal atrophy, brain volume and gray-white matter ratio. Anatomic sequences including: 1) Coronal 3-D volume T1 weighted gradient echo images with effective slice thickness of 1mm. 2) Axial FLAIR (fluid attenuated inversion recovery)
Time Frame: 3 months
Population: All participants with both pre- and post-therapy brain MRI examinations.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) | Matching Placebo Twice a Day (BID)
Number analyzed (Participants) | 7 | 8
Participants
  Functional MRI | 2 | 0
  Structural MRI | 0 | 0

9. Other Pre Specified Outcome: Change in Plasma Cytokines
Description: Mean change plasma cytokines from baseline to post intervention with Cognutrin vs. placebo. Inflammatory markers-Cytokines were measured with a panel including IFN-g, IL-6, IL-8 and INF-alpha.
Time Frame: 3 months
Population: All evaluable participants at time of analysis
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | A - Cognutrin #1 | B - Cognutrin #2 | C - Placebo #1 | D - Placebo #2
Number analyzed (Participants) | 5 | 5 | 9 | 9
pg/mL
  IFN-g | 6.23 (2.3) | 8.3 (2.48) | 6.2 (1.72) | 4.64 (1.85)
  IL-10 | 0.29 (0.07) | 0.2 (0.03) | 0.18 (0.05) | 0.22 (0.03)
  IL-6 | 0.55 (0.21) | 2.07 (1.05) | 1.14 (0.16) | 1.5 (0.78)
  IL-8 | 5.56 (0.92) | 8.55 (2) | 7.82 (0.69) | 8.02 (1.49)
  INF-α | 2.29 (0.19) | 2.53 (0.36) | 2.61 (0.14) | 2.61 (2.61)

ADVERSE EVENTS:
Time Frame: 2 years, 10 months
Arm/Group | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) | Matching Placebo Twice a Day (BID)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 10/18 | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) (N=18) | Matching Placebo Twice a Day (BID) (N=18)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) — Not related to study treatment. Participant was randomized to Treatment Arm but never started study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognutrin (n-3 Fatty Acids + Anthocyanins) Twice a Day (BID) (N=18) | Matching Placebo Twice a Day (BID) (N=18)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolism and nutrition disorders, Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The main reason for not completing baseline or post intervention MRI were: (a) Claustrophobia or fear of being in an MRI and (b) metal bands in breast in preparation for to breast reconstruction that prohibited these participants being in MRI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-10-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT01823991/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT01823991/ICF_001.pdf